CLINICAL TRIAL: NCT01009736
Title: Biomarkers of Prostate and Cardiovascular Health of Men Undergoing Prostatectomy Consuming Different Amounts of Soy-Tomato Juice
Brief Title: Effects of Tomato-Soy Juice on Biomarkers in Patients With Prostate Cancer Undergoing Prostatectomy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Steven Clinton, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-07041; NCI-2012-01373 (Registry Identifier: Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2009-11-06; First posted 2009-11-09 (Estimated); Last update posted 2014-10-16 (Estimated); Status verified 2014-10

CONDITIONS: Prostate Cancer
Keywords: stage I prostate cancer; stage IIB prostate cancer; stage IIA prostate cancer; stage III prostate cancer; stage IV prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Dietary Supplement: tomato-soy juice
Other: laboratory biomarker analysis
Other: pharmacological study
Procedure: therapeutic conventional surgery

SUMMARY:
RATIONALE: Tomato-soy juice may slow the growth of tumor cells. Studying samples of blood and tissue from patients with prostate cancer in the laboratory may help doctors identify biomarkers related to cancer. It may also help doctors understand the effect of tomato-soy juice on biomarkers.

PURPOSE: This phase I/II trial is studying the side effects of tomato-soy juice and its effect on biomarkers in patients with prostate cancer undergoing prostatectomy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the incidence and severity of toxicity associated with tomato-soy juice in patients undergoing prostatectomy.

Secondary

* Quantify changes in the content and distribution of soy isoflavones and tomato phytochemicals (carotenoids and polyphenols) to the prostate and correlate tissue content and patterns with blood and urinary concentrations of these compounds and their metabolites.
* Determine blood hormonal patterns and biomarkers of oxidative stress that favor prostate cancer prevention.
* Investigate histopathologic and molecular biomarkers associated with prostate carcinogenesis that may serve as surrogate endpoint biomarkers and provide information regarding their ability to be modulated by the tomato-soy juice.
* Examine several critical histopathologic endpoints, including systemic hormones, cell/matrix interactions in the tumor microenvironment, and molecular processes within the tumor cells (tumor grade and nuclear morphometry, tumor stage, proliferation index, apoptotic index, and angiogenesis/vascularity).
* Determine if consumption of tomato-soy juice alters molecular markers in the human prostate, including neuroendocrine markers such as IGF-I and IGF-BP3, signal transduction markers such as PTEN (phosphatase and tensin homologue) and phospho-AKT, and angiogenesis regulators such as VEGF (vascular epithelial growth factor).

OUTLINE: Patients receive tomato-soy juice daily for 4 weeks. Patients then undergo prostatectomy.

Patients complete urologic symptom and quality-of-life questionnaires.

Blood, urine, and tissue samples are collected for biomarker and pharmacokinetic analysis.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven carcinoma of the prostate.
* Have chosen radical prostatectomy (or cystoprostatectomy) for treatment of their disease after presented all possible options by medical team.
* Not receiving neoadjuvant hormonal or chemotherapy (other clinical trials)
* ECOG (Eastern Cooperative Oncology Group) performance status 0-1
* Not currently taking lycopene, soy dietary supplements, or "alternative" products (i.e. PC-SPES, Saw Palmetto).
* BUN/Cr (Blood urea nitrogen and serum creatinine), liver enzymes, CBC (complete blood count), and PT/PTT/INR (prothrombin time/partial thromboblastin time) within normal limits.
* Voluntarily agree to participate and a sign an informed consent document.
* Agree to have prostate biopsy blocks provided to the study for evaluation.
* Agree to consume a standardized vitamin and mineral supplement and avoid other nutrition, dietary, or alternative medications/supplements for the duration of the study.

Exclusion:

* Active malignancy other than prostate cancer that requires therapy.
* History of traumatic or surgical castration.
* History of pituitary hormone diseases that currently require supplemental hormonal administration (thyroid hormones, ACTH, growth hormone) or other endocrine disorders requiring hormone administration with the exception of diabetes and osteoporosis.
* Are taking certain medications. No concurrent finasteride (Proscar) or other hormonal agents for chemoprevention/treatment of BPH (benign prostate hyperplasia). Utilizing prescription medications for urinary outlet obstructive symptoms will not be permitted. The use of non-prescription substances to improve urinary tract symptoms will not be permitted (i.e. Saw Palmetto, other herbal, alternative products).
* Have certain medical conditions including: malabsorptive disorders or other metabolic disorders requiring special diet recommendations, severe constipation (may be accentuated by soy), a recent history of anemia or iron deficiency (possible accentuation by soy), or hypertension that requires a strict low sodium diet (tomato juice is high in sodium). The severity of these conditions and eligibility will be defined after careful review of the medical records by Dr. Clinton.
* Have a known allergy to soy or tomato components.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-01; Primary Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of toxicity associated with tomato-soy juice

SECONDARY OUTCOMES:
Changes in the content and distribution of soy isoflavones and tomato phytochemicals (carotenoids and polyphenols) to the prostate and correlation of tissue content and patterns with blood and urinary concentrations of these compounds and their metab ...
Blood hormonal patterns and biomarkers of oxidative stress that favor prostate cancer prevention
Histopathologic and molecular biomarkers associated with prostate carcinogenesis that may serve as surrogate endpoint biomarkers and their ability to be modulated by the tomato-soy juice
Systemic hormones, cell/matrix interactions in the tumor microenvironment, and molecular processes within the tumor cells, including tumor grade and nuclear morphometry, tumor stage, proliferation index, apoptotic index, and angiogenesis/vascularity
Alteration of molecular markers in the human prostate, including neuroendocrine markers such as IGF-I and IGF-BP3, signal transduction markers such as PTEN (phosphatase and tensin homologue) and phospho-AKT, and angiogenesis regulators such as VEGF ( ...

CONTACTS AND LOCATIONS:
Overall Officials: Steven K. Clinton, MD, PhD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Arthur G. James Cancer Hospital and Richard J. Solove Research Institute at Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

REFERENCES:
- [Derived] Moran NE, Thomas-Ahner JM, Fleming JL, McElroy JP, Mehl R, Grainger EM, Riedl KM, Toland AE, Schwartz SJ, Clinton SK. Single Nucleotide Polymorphisms in beta-Carotene Oxygenase 1 are Associated with Plasma Lycopene Responses to a Tomato-Soy Juice Intervention in Men with Prostate Cancer. J Nutr. 2019 Mar 1;149(3):381-397. doi: 10.1093/jn/nxy304. PMID 30801647
- [Derived] Grainger EM, Moran NE, Francis DM, Schwartz SJ, Wan L, Thomas-Ahner J, Kopec RE, Riedl KM, Young GS, Abaza R, Bahnson RR, Clinton SK. A Novel Tomato-Soy Juice Induces a Dose-Response Increase in Urinary and Plasma Phytochemical Biomarkers in Men with Prostate Cancer. J Nutr. 2019 Jan 1;149(1):26-35. doi: 10.1093/jn/nxy232. PMID 30476157
- See also: The Jamesline — http://cancer.osu.edu